CLINICAL TRIAL: NCT05393856
Title: CG-549 Tablet Pharmacokinetics Study: An Open-label, Single Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of a Tablet Formulation of CG-549 in Healthy Subjects
Brief Title: CG-549 Tablet Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CG-549-1-03
Record Dates: First submitted 2019-12-10; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fed state in PART B (Experimental)
  Interventions: Drug: CG-549
- fasted state in PART B (Experimental)
  Interventions: Drug: CG-549

INTERVENTIONS:
Drug: CG-549 — PART A (open-label)
  Period 1: single oral dose. Period 2: After PK evaluation of period 1. Period 3: After PK evaluation of period 2.
  PART B (randomized)
  * Period 1: a single oral dose of ZZ mg CG-549 on Day 1 in fed or fasted state.
  * Period 2: a single oral dose of ZZ mg CG-549 on Day 1 in fasted or fed state.
  Other Names: PART A and PART B

SUMMARY:
This will be an open label, crossover, single dose study consisting of 2 parts (Part A and Part B) in a total of 24 healthy male and female subjects.

DETAILED DESCRIPTION:
Part A Part A is an open-label, 3-period, fixed-sequence, escalating dose study in 6 healthy subjects to find a tablet dose that results in a CG-549 exposure that is expected to be safe and potentially efficacious (i.e., within the targeted efficacious exposure range as defined below).

Subjects will receive the following treatments of the tablet formulation of CG-549, in the fed state:

* Period 1: a single oral dose of 300 mg CG-549 on Day 1.
* Period 2: a single oral dose of XX mg CG-549 on Day 1. After interim PK evaluation of Period 1, the CG-549 dose of Period 2 will aim at reaching the lower end of the targeted efficacious exposure range.
* Period 3: a single oral dose of YY mg CG-549 on Day 1. After interim PK evaluation of Period 2, the CG-549 tablet dose of Period 3 will aim at reaching the higher end of the targeted efficacious exposure range.

Doses XX and YY will be multiples of 300 mg and will not exceed 3 times the dose used in the preceding period.

After interim PK evaluation of all periods in Part A, the CG-549 dose and the type of breakfast to be used in Part B will be selected which is anticipated to result in an exposure that is expected to be safe and potentially efficacious.

Part B Part B is an open-label, 2-period, randomized crossover study in 18 healthy subjects to confirm that the selected dose of the tablet formulation of CG-549 results in a CG-549 exposure that is expected to be safe and potentially efficacious, and to compare the PK profiles of a single dose of the tablet formulation of CG 549 between the fed and the fasted states.

Subjects will receive the following treatments of the tablet formulation of CG-549:

* Period 1: a single oral dose of ZZ mg CG-549 on Day 1 in fed or fasted state.
* Period 2: a single oral dose of ZZ mg CG-549 on Day 1 in fasted or fed state. Dose ZZ will be a multiple of 300 mg.

There will be 2 treatment sequences in the study: fed-fasted and fasted-fed. Subjects will be randomly assigned to a treatment sequence in a 1:1 ratio. In the fed state, subjects will either receive a high-fat or a medium fat breakfast.

ELIGIBILITY:
Key Inclusion Criteria:

1. Sex:Males and females
2. Age:18 to 55 years, inclusive, at screening
3. Weight:≥50 kg, at screening
4. Body mass index:18.0 to 30.0 kg/m2, inclusive, at screening
5. Smoking behavior :Non-smoking or smoking ≤5 cigarettes, 1 cigar, or 1 pipe per day
6. Other criteria:Liver enzymes within the normal range and creatine phosphokinase within 2.0 times the normal range

Key Exclusion Criteria:

1. Previous participation in the current study.
2. Employee of PRA or the Sponsor.
3. History of bacterial or viral infection requiring treatment with antibiotics or antivirals within 1 month prior to screening.
4. Presence or history of esophageal or gastroduodenal ulceration within 1 month prior to screening.
5. Significant and/or acute illness within 5 days prior to the first drug administration that may impact safety assessments, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of CG549 | up to 4 weeks
Area Under the Concentration-Time Curve (AUC) of CG549 | up to 4 weeks

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Velinova, Ph.D, Principal Investigator — PRA Health Sciences (PRA) - Early Development Services (EDS)
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen, Netherlands